CLINICAL TRIAL: NCT00972894
Title: Prospective Evaluation of a Polymerase Chain Reaction (PCR) Assay (GenExpert DX™) for the Rapid Detection of Recto-vaginal Group B Streptococcus (GBS) Colonisation During Intrapartum Screening
Brief Title: Group B Streptococcus (GBS) Polymerase Chain Reaction (PCR) Concordance Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HCA International Limited (Other)
Responsible Party: Dr Bignall, The Portland Hospital
Other Study IDs: CTO/08/024
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2009-09

CONDITIONS: Group B Streptococcus
Keywords: Group B streptococcus; Polymerase chain reaction; PCR; Intrapartum screening; Risk factors; arly onset Group B streptococcus infection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — Vaginal culture swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are comparing three different methods of testing for an infection which is commonly found in women. The infection is caused by a bacterium called Group B Streptococcus. About 10-30% of women carry GBS in the vagina or rectum.

During labour this infection can be passed to the neonate. This can lead to the baby developing a serious infection.

However, research has shown that if antibiotic treatment is given to GBS carrying women during labour most of these infections can be avoided.

A new bedside test known as PCR has been shown to produce a GBS diagnostic result in less than an hour. In clinical trials conducted in the US and France this method has been shown to be more accurate than either prenatal vaginal swabs or risk factor assessment. For this reason, PCR may be helpful in screening and treating GBS positive women in the UK.

In this study the investigators will compare each of the following three methods of diagnosis to a gold standard.

* Prenatal vaginal culture swab (at 35 to 37 weeks gestation)- The US approach.
* Risk factor assessment (at the time of admission for labour)- The UK approach
* The new PCR test (at the time of your labour admission)

The investigators will compare the accuracy of each of these methods with the most accurate method for determining the GBS status during labour. This 'most accurate' method is a highly sensitive swab test which unfortunately takes several days to produce a result. For this reason this test will not tell the investigators whether prophylactic antibiotics may be useful during labour (Receiving them after birth is ineffective).

If PCR is shown to be a more accurate method of identifying GBS positive women this may help to reduce the number of infections in new born infants and as a result may help to save lives.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study if they are;
* 18 years or older
* Pregnant and planned admission to Portland Hospital whether full-term or otherwise.
* Willing and able to give informed consent prenatally.

Exclusion Criteria:

* Scheduled for non vaginal birth

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant females
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bignall, Principal Investigator — Portland Hospital
Locations (2):
- United Kingdom (2):
  - The Portland Women ansd Children's Hospital, London
  - The Portland Hospital, London